CLINICAL TRIAL: NCT00484523
Title: Constitution of a Standardized Neural Imaging Database in Healthy Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2007/09
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: To constitute a standardized database of multimode neural imaging.
MeSH Terms: interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Magnetic Resonance Spectroscopy

INTERVENTIONS:
Procedure: SPET, PET and MRI — 60 healthy subjects after a a consultation with a neurologist for wich 4 examinations will be programmed in two days ( 1 cerebral MRI, 1pet scan, 1 spet, 1 datascan

SUMMARY:
MRI is a powerful imaging tool used for the precise study of brain morphology (morphometric study, tissue study, study of connectivity).

Isotopic examinations by Single Photon Emission Tomography (SPET) and Positron Emission Tomography (PET) are used to explore cerebral perfusion metabolism (99mTc- ECD SPET and 18FDG PET), as well as dopaminergic neurotransmission (123I FP-CIT SPET, DATSCAN®).

These examinations routinely contribute to the clinical diagnosis and surveillance of many neurological pathologies (dementias, Parkinson syndromes, epilepsies, concussions, vascular pathology, brain tumors, etc.).

As a result of the original morphological and functional information they provide, these examinations are being increasingly included in clinical research protocols involving the brain.

The absolute or relative quantification of anomalies observed, however, can be obtained only after comparison to a database of normal subjects.

The creation of these databases is currently limited by their cost and strictly single center nature (physical characteristics of each center's MRI, gamma cameras and PET scanner).

The aim of this multidisciplinary study is to constitute a standardized database of multimode neural imaging (SPET, PET and MRI) to be able to objectively quantify anomalies observed in patients, at the scale of a group or an individual, for the diagnosis and surveillance of neurological diseases.

Participants will be paid €350. 60 healthy subjects between 20 and 80 years of age (30 men and 30 women) will be recruited over 3 years. 4 examinations will be programmed over 2 days (one cerebral MRI, on 18FDG PET, one 99mTc-ECD SPET and one DATSCAN®).

The strictly single center character of this study is explained by the variability of the physical characteristics of the imaging equipment used (MRI, SPET and PET scan) inherent to each center.

ELIGIBILITY:
Inclusion Criteria:

* no neurological or psychiatric history
* no serious disease
* receiving no neurotropic
* no alcoholism
* no drug addiction
* social security cover
* written informed consent

Exclusion Criteria:

* pregnancy
* breast feeding
* contraindication to MRI, SPET or PET exploration

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
precise brain morphology | two days

CONTACTS AND LOCATIONS:
Overall Officials: Eric GUEDJ, AHU, Principal Investigator — Assistance Publique des Hôpitaux de Marseille
Locations (1):
- CHU Timone, Marseille, France

REFERENCES:
- [Derived] Mairal E, Barberon B, Laine N, Coulange M, Guedj E. Reversible widespread brain 18F-FDG PET hypometabolism in chronic fatigue syndrome treated by hyperbaric oxygen therapy. Eur J Nucl Med Mol Imaging. 2021 May;48(5):1680-1681. doi: 10.1007/s00259-020-05122-0. Epub 2021 Jan 9. No abstract available. PMID 33420913
- [Derived] Didic M, Felician O, Gour N, Bernard R, Pecheux C, Mundler O, Ceccaldi M, Guedj E. Rhinal hypometabolism on FDG PET in healthy APO-E4 carriers: impact on memory function and metabolic networks. Eur J Nucl Med Mol Imaging. 2015 Sep;42(10):1512-21. doi: 10.1007/s00259-015-3057-y. Epub 2015 Apr 22. PMID 25900275
- [Derived] Arthuis M, Micoulaud-Franchi JA, Bartolomei F, McGonigal A, Guedj E. Resting cortical PET metabolic changes in psychogenic non-epileptic seizures (PNES). J Neurol Neurosurg Psychiatry. 2015 Oct;86(10):1106-12. doi: 10.1136/jnnp-2014-309390. Epub 2014 Dec 2. PMID 25466258